CLINICAL TRIAL: NCT03578640
Title: The Efficacy of Elbasvir/Grazoprevir Fixed-Dose Combination for 8 Weeks in Treatment-Naïve, Non-Cirrhotic, HCV GT4-Infected Patients: A Single-Center, Single-Arm, Open-Label, Phase III Trial
Brief Title: Eight Weeks of Elbasvir/Grazoprevir in the Treatment of HCV Genotype 4
Acronym: ELEGANT-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Ahmad A AlEid, MD, Staff Physician, Department of Gastroenterology and Hepatology, Consultant Advanced Hepatology and Liver Transplantation, Principal Investigator of the ELEGANT-4 trial, King Fahad Medical City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-226
Record Dates: First submitted 2018-06-06; First posted 2018-07-06 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C Virus; Chronic Hepatitis C; Genotype 4; Treatment-naive; Non-cirrhotic
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — elbasvir; grazoprevir; Tablets; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Intervention Model Description: An interventional, single-center, single-arm study among 30 patients who are treatment naïve, have no advanced fibrosis and mono-infected with HCV-GT4.
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Elbasvir, Grazoprevir 50-100Mg Oral Tablet
  Interventions: Drug: Elbasvir, Grazoprevir 50-100Mg Oral Tablet

INTERVENTIONS:
Drug: Elbasvir, Grazoprevir 50-100Mg Oral Tablet — Daily, fixed-dose combination of Elbasvir 50 mg and Grazoprevir 100 mg given in a single oral tablet for 8 weeks.
  Other Names: Elbasvir / Grazoprevir Oral Tablet (Zepatier)

SUMMARY:
To evaluate the safety and efficacy of a daily, fixed-dose, 8-week course combination of Elbasvir/Grazoprevir in treatment-naïve, non-cirrhotic patients who are mono-infected with hepatitis C, genotype 4.

DETAILED DESCRIPTION:
The treatment of hepatitis C has gone through significant advances in the last few years with the development of direct-acting antivirals "DAAs." Since 2013, many DAAs have been approved for the treatment of HCV with excellent efficacy and safety profiles. The major hurdle in treating patients on a large scale is the high cost of the current treatment regimens. Multiple approaches have been proposed, among them, a shortened treatment regimen of 6 to 8 weeks rather than the standard 12-week-regimen. The strategy of shortening the treatment will help in reducing the cost by 33% to 50%. Thus, it will increase the availability of the treatment to more patients.

Zepatier is a combination drug of Elbasvir (EBR), an NS5A inhibitor, and Grazoprevir (GZR), a potent NS3/4A inhibitor. This study is being proposed to address two main issues. First, collecting information on the safety and efficacy of a shortened course of zepatier (8 weeks instead of the standard 12 weeks) in patients who are treatment-naïve, non-cirrhotic and mono-infected with HCV. Second, to investigate whether this course provides similar clinical outcomes to the standard regimen in HCV-Genotype 4, which is the most common genotype in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Chronically infected with HCV genotype 4.
3. Treatment naïve.
4. No advanced fibrosis. Defined by the absence of clinical, radiological and laboratory signs of cirrhosis, and fibrosis assessment consistent with fibrosis stage (Metavir F2) or less by liver biopsy or transient elastography.
5. Not expected to leave the country for six months after the end of the intervention.

Exclusion Criteria:

1. Incapability of providing an informed consent to participate in the study.
2. Advanced fibrosis (Metavir F3) or cirrhosis (Metavir F4).
3. HIV or HBV co-infection
4. Organ transplant recipients.
5. Type 2 or 3 cryoglobulinemia with end-organ manifestations.
6. Proteinuria, nephrotic syndrome, or membranoproliferative glomerulonephritis
7. Patients with a higher risk of transmitting the disease (Dialysis patients, incarcerated individuals, and intravenous drug abusers).
8. The use of any medication that has major interactions with Elbasvir or Grazoprevir as defined by the University of Liverpool drug interaction database, and cannot be discontinued or replaced with other alternatives.
9. Pregnancy.
10. History of hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after the end of intervention (SVR-12). | At 12 weeks after the end of intervention.
  Viral RNA below the level of detection at 12 weeks after the end of the intervention.
  (Hepatitis C viral load evaluated by polymerase chain reaction (PCR) with a cutoff of 20 IU/mL for detectability.)

SECONDARY OUTCOMES:
Sustained virological response at 4 weeks after the end of intervention (SVR-4). | At 4 weeks after the end of intervention.
  Hepatitis C viral RNA below the level of detection at 4 weeks after the end of the intervention.
Serious and treatment-related adverse events. | From the first day of intervention until the end of week 4 after the intervention is finished.
  Number of patients with serious and treatment-related adverse events based on the common terminology criteria (CTCAE 4.03), or death during the follow-up period.
Changes in the quality of life: Hepatitis Quality of Life Questionnaire (HQLQ) | Quality of life evaluations will take place over three occasions. The first will be at baseline (upon treatment initiation), the second will be during treatment/at the end of treatment, and the last will be 12 weeks after the end of treatment
  To assess this outcome, a self-administered questionnaire called the "Hepatitis Quality of Life Questionnaire" (HQLQ) will be used. The HQLQ is composed of 7 domains; the physical and mental components (PCS and MCS, respectively), a self-evaluated health transition item (SET), and four hepatitis-related items. The latter include general health distress (HD), psychological well-being (PWB), hepatitis-specific functional limitations (HLIM), and hepatitis-specific health distress (HHD) sub-scales. Higher numbers on each component/scale represent better results (e.g., better physical, emotional, and psychological functioning, and little to no limitations in these aspects). Higher scores on the self-evaluated transition item, however, represent less favorable results.
  These assessments will take place over three occasions. The first will be upon initiating the treatment, the second will be during/by the end of treatment, and the last will take place 12 weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahad Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Serfaty L, Zeuzem S, Vierling JM, et al. High efficacy of the combination HCV regimen grazoprevir and elbasvir for 8 or 12 weeks with or without ribavirin in treatment-naive, noncirrhotic HCV GT1b-infected patients: an integrated analysis. Program and abstracts of the 2015 Annual Meeting of the American Association for the Study of Liver Diseases; November 13-17, 2015; San Francisco, California. Abstract 701.
- [Result] STREAGER Interim Analysis: High Rate of SVR With 8 Weeks of Elbasvir/Grazoprevir in Treatment-Naive Patients With Genotype 1b HCV Infection and F0-F2 Fibrosis; 2017 Annual Meeting of the American Association for the Study of Liver Diseases; Washington DC; Posted online October 27, 2017.
- [Result] Lawitz E, Poordad F, Gutierrez JA, Wells JT, Landaverde CE, Evans B, Howe A, Huang HC, Li JJ, Hwang P, Dutko FJ, Robertson M, Wahl J, Barr E, Haber B. Short-duration treatment with elbasvir/grazoprevir and sofosbuvir for hepatitis C: A randomized trial. Hepatology. 2017 Feb;65(2):439-450. doi: 10.1002/hep.28877. Epub 2016 Dec 19. PMID 27770561
- [Result] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518
- [Derived] AlEid A, Al Balkhi A, Qutub A, Abbarh S, AlLehibi A, Almtawa A, Al Otaibi N, AlGhamdi A, AlGhamdi A, Alamr A, Ahmad S, Al Sayari K, Al Ibrahim B, AlKhathlan A. The efficacy of Elbasvir/Grazoprevir fixed-dose combination for 8 weeks in HCV treatment and health-related quality of life (HRQoL) in treatment-naive, non-cirrhotic, genotype 4-infected patients (ELEGANT-4): A single-center, single-arm, open-label, phase 3 trial. Saudi J Gastroenterol. 2022 May-Jun;28(3):225-232. doi: 10.4103/sjg.sjg_374_21. PMID 35142658
- See also: C-WORTHY trial — http://www.natap.org/2015/AASLD/AASLD_169.htm
- See also: Short-duration treatment with elbasvir/grazoprevir and sofosbuvir for hepatitis C: A randomized trial. Hepatology. 2017 Feb;65(2):439-450. doi: 10.1002/hep.28877. Epub 2016 Dec 19. — https://www.ncbi.nlm.nih.gov/pubmed/27770561
- See also: Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. — https://www.ncbi.nlm.nih.gov/pubmed/28193518